CLINICAL TRIAL: NCT05821803
Title: The Effect of Exercise Training and Arch Supported Insoles on Balance and Vertical Jump Performance in Football Players With Foot Pronation Deformity: Randomized Controlled Trial
Brief Title: The Effect of Exercise Training and Arch Supported Insoles on Balance and Vertical Jump Performance in Football Players With Foot Pronation Deformity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: FootBalance (Unknown)
Responsible Party: Principal Investigator, Gizem Karadeniz, Physiotherapist, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GizemK
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Foot; Pronation, Congenital
Keywords: Foot pronation; Insoles; Footcore exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Insoles
  Foot Core Exercises
  Interventions: Other: Using Insoles; Other: Foot Core Exercises
- Control Group (Active Comparator): Insoles
  Interventions: Other: Using Insoles

INTERVENTIONS:
Other: Using Insoles — FootBalance %100 Control Orthopedic insoles used for 4 weeks.
Other: Foot Core Exercises — 4 weeks including
  Arms: Experimental Group

SUMMARY:
This study aims to investigate the effects of foot pronation exercises and arch support insoles on balance and vertical jump test in football players.

DETAILED DESCRIPTION:
The study took place in FootBalance Turkey, which works on foot analysis and insoles.

30 professional football players with pronation who divided into two groups. The football players in the Experimental Group used insoles and also participated the foot core exercise program twice a week for 4 weeks duration. The football players in the Control Group just used the insoles.We used the FootBalance assessmnet system for insoles. Navicular Drop Test, Y Balance Test, Flamingo Testand Vertical Jump Test applied to evalute foot pronation, dynamic balance, static balance and jump performace respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in research
2. To be between the ages of 18-45
3. Overpronation foot ( navicular drop test over 10 mm and FootBalance device with visual display)
4. Professional football players at least 5 years

Exclusion Criteria:

1. History of surgery for musculoskeletal structures in both lower extremities
2. History of fracture in both lower extremities
3. Acute injury of the musculoskeletal structures of other joints of the lower extremity affecting joint function and integrity in the last 3 months
4. Have any other knee pathology
5. Balance or vestibular disorder

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Navicular Drop Test | 4 weeks
  It is the one of the static foot assessment tool and is intended to represent the sagittal plane displacement of the navicular tuberosity from a neutral position.
Y Balance Test/ Dynamic Balance Evaluation | 4 weeks
  The Star Excursion Balance Test (SEBT) is a dynamic test that requires strength, flexibility, and proprioception. It is a measure of dynamic balance that provides a significant challenge to athletes and physically active individuals.
Flamingo Balance Test/ Static Balance Evalutaion | 4 weeks
  The flamingo balance test is a total body balance test in order to test static balance.
Vertical Jump Test | 4 weeks
  Vertical jump test to determine an athlete's physical ability. The vertical jump as a test of lower body explosive power

CONTACTS AND LOCATIONS:
Locations (1):
- FootBalance Merkez, Istanbul, Şişli, Turkey (Türkiye)